CLINICAL TRIAL: NCT04022018
Title: Study on Adaptive Radiotherapy and Multimodal Information of Cervical Cancer Assisted by Artificial Intelligence
Acronym: SOARAMIOCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong-Shenzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hkuszh2019119
Record Dates: First submitted 2019-07-01; First posted 2019-07-16 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Cervical Cancer; Radiotherapy Side Effect; Biomarker; Artificial Intelligence
Keywords: cervical cancer; adaptive radiotherapy; side effects
MeSH Terms: conditions — Uterine Cervical Neoplasms; Radiation Injuries

STUDY DESIGN:
Intervention Model Description: Total 122 cases of IB2-IVA cervical cancer will be randomly enrolled. Concurrent external volumetric rotational intensity modulated radiotherapy and chemotherapy followed by image-guided adaptive brachytherapy is the treatment strategies of control group patients.
  Concurrent adaptive external volumetric rotational intensity modulated radiotherapy and chemotherapy followed by image-guided adaptive brachytherapy is the treatment strategies of experimental group patients. CT repositioning will be performed after 15fractions of external radiotherapy, then new target volume will be contoured and new radiotherapy plan will be formulated with the assistance of artificial intelligence program. New radiotherapy plan will be performed from the 17th fraction external radiotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adaptive radiotherapy group (Experimental): Concurrent adaptive external volumetric rotational intensity modulated radiotherapy and chemotherapy followed by image-guided adaptive brachytherapy is the treatment strategies of adaptive radiotherapy group patients. CT repositioning will be performed after 15fractions of external radiotherapy, then new target volume will be contoured and new radiotherapy plan will be formulated with the assistance of artificial intelligence program. New radiotherapy plan will be performed from the 17th fraction external radiotherapy.
  Interventions: Radiation: Adaptive radiotherapy
- Control group (Active Comparator): Concurrent external volumetric rotational intensity modulated radiotherapy and chemotherapy followed by image-guided adaptive brachytherapy is the treatment strategies of control group patients.
  Interventions: Radiation: no adaptive radiotherapy

INTERVENTIONS:
Radiation: Adaptive radiotherapy — CT repositioning will be performed after 15fractions of external radiotherapy, then new target volume will be contoured and new radiotherapy plan will be formulated with the assistance of artificial intelligence program. New radiotherapy plan will be performed from the 17th fraction external radiotherapy.
  Arms: Adaptive radiotherapy group
Radiation: no adaptive radiotherapy — Concurrent external volumetric rotational intensity modulated radiotherapy and chemotherapy followed by image-guided adaptive brachytherapy is the treatment strategies of control group patients
  Arms: Control group

SUMMARY:
The standard treatment for non-operative cervical cancer is concurrent external radiation therapy and chemotherapy followed by brachytherapy. During the period of radiotherapy, organ movement and tumor shrinkage may lead to insufficient or excessive radiation dose for the tumor and organs at risk. Adaptive radiotherapy can use images information acquired during treatment as feedback to reduce errors.

Total 122 cases of cervical cancer with stage IB2-IVA will be randomly enrolled. Concurrent external volumetric rotational intensity modulated radiotherapy and chemotherapy followed by image-guided adaptive brachytherapy is the treatment strategies of control group patients.

Concurrent adaptive external volumetric rotational intensity modulated radiotherapy and chemotherapy followed by image-guided adaptive brachytherapy is the treatment strategies of experimental group patients. CT repositioning will be performed after 15fractions of external radiotherapy, then new target volume will be contoured and new radiotherapy plan will be formulated with the assistance of artificial intelligence program. New radiotherapy plan will be performed from the 17th fraction external radiotherapy. Information on side effects, survival, dosimetry, imaging, clinical features, and cost-effectiveness will be collected. The statistical analysis is as follows, First is the difference in grade 3 side effects between the two groups. Second is 2-year PFS and OS differences between the two groups. Third is relationship between dosimetric differences and prognosis. Fourth one is to analyze the prognostic and predictive factors of adaptive radiotherapy from the patient's clinical characteristics, Positron emission tomography-computed tomography(PET/CT), Magnetic Resonance Imaging(MRI) and other multimodal information. Fifth is cost-benefit analysis of Artificial Intelligence(AI).

DETAILED DESCRIPTION:
1. Introduction and background The standard treatment for non-operative cervical cancer is concurrent external radiation therapy and chemotherapy followed by brachytherapy. During the period of radiotherapy, organ movement and tumor shrinkage may lead to insufficient or excessive radiation dose for the tumor and organs at risk. Adaptive radiotherapy can use images information acquired during treatment as feedback to reduce errors.
2. Hypothesis and purpose Main endpoint: adaptive radiotherapy can reduce level 3 side effects or not. Secondary endpoint: 1. The differences of 2-year progression-free survival and overall survival between two groups. 2. To analyze Physical dosimetry differences between two groups, and the correlation between physical dosimetry differences and prognosis also will be evaluated. 3. To analyze the prediction and prognostic factors of adaptive radiotherapy for cervical cancer, and to provide supporting data for the subsequent optimization of cervical cancer treatment. 4. To evaluate the effectiveness of AI and conduct cost-benefit analysis.
3. Trial methodology and design Total 122 cases of IB2-IVA cervical cancer will be randomly enrolled. Concurrent external volumetric rotational intensity modulated radiotherapy and chemotherapy followed by image-guided adaptive brachytherapy is the treatment strategies of control group patients.

   Concurrent adaptive external volumetric rotational intensity modulated radiotherapy and chemotherapy followed by image-guided adaptive brachytherapy is the treatment strategies of experimental group patients. CT repositioning will be performed after 15fractions of external radiotherapy, then new target volume will be contoured and new radiotherapy plan will be formulated with the assistance of artificial intelligence program. New radiotherapy plan will be performed from the 17th fraction external radiotherapy.

   Meanwhile, concurrent chemotherapy regimen is cisplatin 40mg/m2/week (the maximum weekly dose should less than or equal to 70mg and no more than 6cycles). Information on side effects, survival, dosimetry, imaging, clinical features, and cost-effectiveness will be collected. The statistical analysis is as follows, First is the difference in grade 3 side effects between the two groups. Second is 2-year PFS and OS differences between the two groups. Third is relationship between dosimetric differences and prognosis. Fourth one is to analyze the prognostic and predictive factors of adaptive radiotherapy from the patient's clinical characteristics, PET/CT, MRI and other multimodal information. Fifth is cost-benefit analysis of AI.
4. Anticipated result and potential impact Adaptive radiotherapy can reduce side effects and obtain prognosis and prognostic factors of adaptive radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. pathologically confirmed cervical squamous cell carcinoma or adenocarcinoma without treatment before;
2. Age: ≥18 years old;
3. The International Federation of Gynecology and Obstetrics(FIGO) stage: IB2 to IVA, or IVB with only para-aortic lymph node metastasis, refused or could not be treated by surgery;
4. Eastern Cooperative Oncology Group(ECOG)score ≤2;
5. good bone marrow, hematopoietic and liver and kidney function: absolute neutrophil count (ANC) ≥ 1.5 ☓ 109 / L, the platelet count ≥100 ☓ 109 / L, or hemoglobin > 90 g/L, serum bilirubin < 1.5 ☓ upper limit of normal reference value(ULN), aspartate aminotransferase(AST) and alanine aminotransferase(ALT)< 2.5 ☓ ULN, serum creatinine clearance ≥ 50 ml/min.
6. provide informed consent.

Exclusion Criteria:

1. women in pregnancy or nursing;
2. contraindications to chemoradiotherapy;
3. subjects participating in other clinical trials or participating in other clinical trials within 30 days;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2019-12-18 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
the difference in grade 3 side effects between the two groups | The acute radiotherapy reaction occur from the first day to 90 days after the end of radiotherapy, and the late radiotherapy reaction occur 90 days after radiotherapy.
  Hematologic toxicity, bladder and rectal radiotherapy toxicity were recorded according to the evaluation criteria of common adverse events (CTCAE version 4.03).

SECONDARY OUTCOMES:
2-year PFS differences between the two groups | 2-year PFS
  Follow-up every 3 months within 2 years after the end of radiotherapy, and every 6 months after 2 years. 2-year progression-free survival (PFS) will be calculated.
2-year OS differences between the two groups | 2-year OS
  Follow-up every 3 months within 2 years after the end of radiotherapy, and every 6 months after 2 years. 2-year overall survival (OS) will be calculated.
the correlation between physical dosimetry differences and prognosis | correlation between physical dosimetry differences and 2year PFS
  To analyze Physical dosimetry differences between two groups, and the correlation between physical dosimetry differences and prognosis also will be evaluated.
the predictive factors for the response rate of concurrent chemoradiotherapy for cervical cancer | 3 months after radiotherapy
  To investigate the predictive factors for the response rate of concurrent chemoradiotherapy for cervical cancer. The investigating multimodal factors include patients'demographic characteristics, ECOG score, disease staging, human papilloma virus(HPV) status, tumor standard uptake value (SUV) of PET/CT and tumor apparent diffusion coefficient (ADC) value of MRI, squamous cell carcinoma antigen, lymphocyte and hemoglobin. Response rate is assessed at 3 months after completion of radiotherapy by MRI according to RECIST 1.1 criteria.
the prognostic factors for the 2-year overall survival rate of patients with cervical cancer after concurrent chemoradiotherapy | 2 years after radiotherapy
  To investigate the prognostic factors for the 2-year overall survival rate of patients with cervical cancer after concurrent chemoradiotherapy. The investigating multimodal factors include patients'demographic characteristics, ECOG score, disease staging, human papilloma virus(HPV) status, tumor standard uptake value (SUV) of PET/CT and tumor apparent diffusion coefficient(ADC) value of MRI, squamous cell carcinoma antigen, lymphocyte and hemoglobin. Overall survival is calculated from the date of diagnosis of cervical cancer to the date of death from any cause.
the time difference between labor and an artificial intelligence to design radiotherapy plans | 2years
  Compare the efficiency AI and labor.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Yuan Xu, master, Principal Investigator — HongKong University Shenzhen Hospital
Locations (1):
- HongKong University Shenzhen Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
The results will be published as papers, but the original data will not be Shared

REFERENCES:
- [Background] Arbyn M, Castellsague X, de Sanjose S, Bruni L, Saraiya M, Bray F, Ferlay J. Worldwide burden of cervical cancer in 2008. Ann Oncol. 2011 Dec;22(12):2675-2686. doi: 10.1093/annonc/mdr015. Epub 2011 Apr 6. PMID 21471563
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Kjaer SK, Frederiksen K, Munk C, Iftner T. Long-term absolute risk of cervical intraepithelial neoplasia grade 3 or worse following human papillomavirus infection: role of persistence. J Natl Cancer Inst. 2010 Oct 6;102(19):1478-88. doi: 10.1093/jnci/djq356. Epub 2010 Sep 14. PMID 20841605
- [Background] Parkin DM, Bray F, Ferlay J, Pisani P. Global cancer statistics, 2002. CA Cancer J Clin. 2005 Mar-Apr;55(2):74-108. doi: 10.3322/canjclin.55.2.74. PMID 15761078
- [Background] International Collaboration of Epidemiological Studies of Cervical Cancer. Comparison of risk factors for invasive squamous cell carcinoma and adenocarcinoma of the cervix: collaborative reanalysis of individual data on 8,097 women with squamous cell carcinoma and 1,374 women with adenocarcinoma from 12 epidemiological studies. Int J Cancer. 2007 Feb 15;120(4):885-91. doi: 10.1002/ijc.22357. PMID 17131323
- [Background] Dugue PA, Rebolj M, Garred P, Lynge E. Immunosuppression and risk of cervical cancer. Expert Rev Anticancer Ther. 2013 Jan;13(1):29-42. doi: 10.1586/era.12.159. PMID 23259425
- [Background] Barnholtz-Sloan J, Patel N, Rollison D, Kortepeter K, MacKinnon J, Giuliano A. Incidence trends of invasive cervical cancer in the United States by combined race and ethnicity. Cancer Causes Control. 2009 Sep;20(7):1129-38. doi: 10.1007/s10552-009-9317-z. Epub 2009 Mar 1. PMID 19253025
- [Background] Rose PG, Bundy BN, Watkins EB, Thigpen JT, Deppe G, Maiman MA, Clarke-Pearson DL, Insalaco S. Concurrent cisplatin-based radiotherapy and chemotherapy for locally advanced cervical cancer. N Engl J Med. 1999 Apr 15;340(15):1144-53. doi: 10.1056/NEJM199904153401502. PMID 10202165
- [Background] Chemoradiotherapy for Cervical Cancer Meta-Analysis Collaboration. Reducing uncertainties about the effects of chemoradiotherapy for cervical cancer: a systematic review and meta-analysis of individual patient data from 18 randomized trials. J Clin Oncol. 2008 Dec 10;26(35):5802-12. doi: 10.1200/JCO.2008.16.4368. Epub 2008 Nov 10. PMID 19001332
- [Background] Klopp AH, Moughan J, Portelance L, Miller BE, Salehpour MR, Hildebrandt E, Nuanjing J, D'Souza D, Souhami L, Small W Jr, Gaur R, Jhingran A. Hematologic toxicity in RTOG 0418: a phase 2 study of postoperative IMRT for gynecologic cancer. Int J Radiat Oncol Biol Phys. 2013 May 1;86(1):83-90. doi: 10.1016/j.ijrobp.2013.01.017. PMID 23582248
- [Background] Tyagi N, Lewis JH, Yashar CM, Vo D, Jiang SB, Mundt AJ, Mell LK. Daily online cone beam computed tomography to assess interfractional motion in patients with intact cervical cancer. Int J Radiat Oncol Biol Phys. 2011 May 1;80(1):273-80. doi: 10.1016/j.ijrobp.2010.06.003. Epub 2010 Nov 23. PMID 21109360
- [Background] Pathy S, Kumar L, Pandey RM, Upadhyay A, Roy S, Dadhwal V, Madan R, Chander S. Impact of Treatment Time on Chemoradiotherapy in Locally Advanced Cervical Carcinoma. Asian Pac J Cancer Prev. 2015;16(12):5075-9. doi: 10.7314/apjcp.2015.16.12.5075. PMID 26163644
- [Background] Perez CA, Grigsby PW, Castro-Vita H, Lockett MA. Carcinoma of the uterine cervix. I. Impact of prolongation of overall treatment time and timing of brachytherapy on outcome of radiation therapy. Int J Radiat Oncol Biol Phys. 1995 Jul 30;32(5):1275-88. doi: 10.1016/0360-3016(95)00220-S. PMID 7635767
- [Background] Petereit DG, Sarkaria JN, Chappell R, Fowler JF, Hartmann TJ, Kinsella TJ, Stitt JA, Thomadsen BR, Buchler DA. The adverse effect of treatment prolongation in cervical carcinoma. Int J Radiat Oncol Biol Phys. 1995 Jul 30;32(5):1301-7. doi: 10.1016/0360-3016(94)00635-X. PMID 7635769
- [Background] Holschneider CH, Petereit DG, Chu C, Hsu IC, Ioffe YJ, Klopp AH, Pothuri B, Chen LM, Yashar C. Brachytherapy: A critical component of primary radiation therapy for cervical cancer: From the Society of Gynecologic Oncology (SGO) and the American Brachytherapy Society (ABS). Brachytherapy. 2019 Mar-Apr;18(2):123-132. doi: 10.1016/j.brachy.2018.11.009. Epub 2019 Jan 18. PMID 30665713
- [Background] Tsien C, Cao Y, Chenevert T. Clinical applications for diffusion magnetic resonance imaging in radiotherapy. Semin Radiat Oncol. 2014 Jul;24(3):218-26. doi: 10.1016/j.semradonc.2014.02.004. PMID 24931097
- [Background] Ohkubo Y, Ohno T, Noda SE, Kubo N, Nakagawa A, Kawahara M, Abe T, Kiyohara H, Wakatsuki M, Nakano T. Interfractional change of high-risk CTV D90 during image-guided brachytherapy for uterine cervical cancer. J Radiat Res. 2013 Nov 1;54(6):1138-45. doi: 10.1093/jrr/rrt073. Epub 2013 Jun 3. PMID 23732770
- [Background] Fu ZZ, Peng Y, Cao LY, Chen YS, Li K, Fu BH. Value of apparent diffusion coefficient (ADC) in assessing radiotherapy and chemotherapy success in cervical cancer. Magn Reson Imaging. 2015 Jun;33(5):516-24. doi: 10.1016/j.mri.2015.02.002. Epub 2015 Feb 7. PMID 25660642
- [Background] Onal C, Yildirim BA, Guler OC, Mertsoylu H. The Utility of Pretreatment and Posttreatment Lymphopenia in Cervical Squamous Cell Carcinoma Patients Treated With Definitive Chemoradiotherapy. Int J Gynecol Cancer. 2018 Oct;28(8):1553-1559. doi: 10.1097/IGC.0000000000001345. PMID 30247248
- [Background] Joo J, Shin HJ, Park B, Park SY, Yoo CW, Yoon KA, Kong SY, Kim YJ, Kim SS, Kim JY. Integration Pattern of Human Papillomavirus Is a Strong Prognostic Factor for Disease-Free Survival After Radiation Therapy in Cervical Cancer Patients. Int J Radiat Oncol Biol Phys. 2017 Jul 1;98(3):654-661. doi: 10.1016/j.ijrobp.2017.02.226. Epub 2017 Apr 13. PMID 28581408
- [Background] Harry VN, Semple SI, Gilbert FJ, Parkin DE. Diffusion-weighted magnetic resonance imaging in the early detection of response to chemoradiation in cervical cancer. Gynecol Oncol. 2008 Nov;111(2):213-20. doi: 10.1016/j.ygyno.2008.07.048. Epub 2008 Sep 6. PMID 18774597
- [Background] Escande A, Haie-Meder C, Maroun P, Gouy S, Mazeron R, Leroy T, Bentivegna E, Morice P, Deutsch E, Chargari C. Neutrophilia in locally advanced cervical cancer: A novel biomarker for image-guided adaptive brachytherapy? Oncotarget. 2016 Nov 15;7(46):74886-74894. doi: 10.18632/oncotarget.12440. PMID 27713124
- [Background] Reuze S, Orlhac F, Chargari C, Nioche C, Limkin E, Riet F, Escande A, Haie-Meder C, Dercle L, Gouy S, Buvat I, Deutsch E, Robert C. Prediction of cervical cancer recurrence using textural features extracted from 18F-FDG PET images acquired with different scanners. Oncotarget. 2017 Jun 27;8(26):43169-43179. doi: 10.18632/oncotarget.17856. PMID 28574816
- [Background] Schernberg A, Bockel S, Annede P, Fumagalli I, Escande A, Mignot F, Kissel M, Morice P, Bentivegna E, Gouy S, Deutsch E, Haie-Meder C, Chargari C. Tumor Shrinkage During Chemoradiation in Locally Advanced Cervical Cancer Patients: Prognostic Significance, and Impact for Image-Guided Adaptive Brachytherapy. Int J Radiat Oncol Biol Phys. 2018 Oct 1;102(2):362-372. doi: 10.1016/j.ijrobp.2018.06.014. Epub 2018 Jun 18. PMID 29920324
- See also: National Comprehensive Cancer Network(NCCN) — https://www.nccn.org/professionals/physician_gls/pdf/cervical.pdf